CLINICAL TRIAL: NCT00136890
Title: The Impact of Positron Emission Tomography (PET) Imaging in Staging Potentially Surgically Resectable Non-small Cell Lung Cancers: A Prospective Multicentre Randomized Clinical Trial
Brief Title: PET Imaging in Potentially Surgically Resectable Non-small Cell Lung Cancers
Acronym: ELPET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CTA-Control-088145
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Non-small-cell Lung Carcinoma
Keywords: Positron-Emission Tomography; PET Scan; Lung Cancer; Thoracic Surgery; Diagnostic; Randomized Controlled Trial; Oncology
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Disease; Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Conventional Staging
- 2 (Experimental): PET Imaging
  Interventions: Procedure: PET Imaging

INTERVENTIONS:
Procedure: PET Imaging — Patients randomized to PET staging will undergo FDG-PET or PET-CT as well as some form of cranial imaging (CT or MRI)
  Arms: 2

SUMMARY:
Lung cancer remains the leading cause of cancer deaths in men and women. Although overall survival remains poor, early stage non-small cell lung cancer (NSCLC) is potentially curable. Improved staging has led to stage-specific therapies such that patients with early stage NSCLC are potential candidates for surgical resection, and those with more advanced disease are spared the morbidity and risk of mortality from thoracotomy and pulmonary resection. Despite contemporary staging techniques, 25-50% of patients who appear to have limited disease amenable to surgical resection go on to die from metastatic lung cancer. If occult micro-metastatic disease that becomes evident later could be detected reliably during the pre-operative assessment, patients harboring such disease could be spared a non-curative thoracotomy. PET imaging has the potential to detect mediastinal and extrathoracic metastatic disease not detected by conventional imaging modalities.

This prospective, multicenter trial will enroll patients with biopsy-proven clinical stage I-IIIA NSCLC who are considered to be candidates for surgical resection with curative intent. Preoperatively, patients will be randomized to conventional staging for metastatic disease (CT liver/adrenals, total body bone scan, and CT with contrast or MRI with gadolinium of the brain) versus whole body PET or PET-CT and brain CT or MRI with contrast/gadolinium.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proof of NSCLC
* Stage I, II, or IIIA NSCLC based upon clinical staging
* The primary lesion appears technically appropriate for surgical resection, based on information from the chest x-ray (CXR) and CT thorax.
* Age over 18 years

Exclusion Criteria:

* Poor pulmonary function precluding radical surgery (inadequate pulmonary reserve for radical surgery) with predicted post-resection forced expiratory volume in 1 second (FEV1) < 0.8 liter or < 40% predicted, and diffusing capacity of the lung for carbon monoxide (DLCO) < 40% predicted
* Poor performance status (Eastern Cooperative Oncology Group [ECOG] 3-4)
* Significant concurrent medical problems (e.g. uncontrolled diabetes, active cardiac problems, significant chronic obstructive pulmonary disease) making the patient unfit for surgery
* Pregnant or lactating females
* Unable to lie supine for imaging with PET
* Patients with previously treated cancer other than non-melanotic skin cancer or carcinoma in situ of the cervix, unless disease-free for 5 years or greater
* Patients who, at the time of the initial evaluation, have already undergone a whole body PET/PET-CT, CT brain, MRI brain, total body bone scan or mediastinoscopy within 8 weeks prior to randomization will be excluded. However, patients who have had a CT scan of the thorax with abdomen are not excluded.
* Failure to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2004-07; Primary Completion 2008-11 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Patients correctly upstaged by PET versus conventional staging | November 2007

SECONDARY OUTCOMES:
Patients erroneously understaged by PET versus conventional staging | November 2008
Overall survival | August 2012
Prognostic ability of PET standard uptake value | August 2011
Sensitivity and specificity of PET in the mediastinum | November 2008
Cost-effectiveness of using PET versus conventional staging | August 2012

CONTACTS AND LOCATIONS:
Overall Officials: Donna E Maziak, MD, Study Chair — The Ottawa Hospital; Gail E Darling, MD, Study Chair — Toronto General Hospital; Mark N Levine, MD, Principal Investigator — Ontario Clinical Oncology Group (OCOG); William Evans, MD, Principal Investigator — Juravinski Cancer Centre
Locations (8):
- Canada (8):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Credit Valley, Mississauga, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Scarborough Hospital, Scarborough Village, Ontario
  - Sunnybrook/TEGH, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - St. Joseph's Health Care, Toronto, Ontario

REFERENCES:
- [Derived] Maziak DE, Darling GE, Inculet RI, Gulenchyn KY, Driedger AA, Ung YC, Miller JD, Gu CS, Cline KJ, Evans WK, Levine MN. Positron emission tomography in staging early lung cancer: a randomized trial. Ann Intern Med. 2009 Aug 18;151(4):221-8, W-48. doi: 10.7326/0003-4819-151-4-200908180-00132. Epub 2009 Jul 6. PMID 19581636